CLINICAL TRIAL: NCT07302399
Title: Comparison of the Postoperative Analgesic Efficacy of SAP and SPSIP Blocks in Patients Undergoing Mammoplasty
Acronym: SPSIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: Karabuk Training and Research Hospital (Other); Çam Sakura Şehir Hastanesi (Unknown); Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ilker Ital, Ass. Prof. Dr, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AIBU-TF-AR-II-005; AIBU-TF-AR-II-005 (Registry Identifier: SPSIP)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Postsurgical Pain; Breast Pain
Keywords: Mammoplasty; Postoperative Pain; SPSIP Block; SAP Block
MeSH Terms: conditions — Pain, Postoperative; Mastodynia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPB Group (Active Comparator): Serratus Anterior Plane Group Drug: 0,25% Bupivacaine 0,5ml/kg (max.20ml) will be used for blocks for each side.
  Interventions: Procedure: Serratus Anterior Plane Block
- SPSIPB Group (Experimental): Serratus Posterior Superior Intercostal Plane Block Group Drug: 0,25% Bupivacaine 0,5ml/kg (max.20ml) will be used for blocks for each side.
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — Application of ultrasound-guided serratus anterior plane block for perioperative analgesia for mammoplasty operations. Serratus anterior plane block will be administered under general anesthesia before the surgery
  Drug: Bupivacaine (Block Drug)
  For block performances, 0,25% Bupivacaine will be used at 0,5 ml/kg (max. 20cc) for each side.
  Other Names: SAP Block
  Arms: SAPB Group
Procedure: Serratus Posterior Superior Intercostal Plane Block — Application of ultrasound-guided serratus anterior plane block for perioperative analgesia for mammoplasty operations. Serratus posterior superior intercostal plane block will be administered under general anesthesia before the surgery
  Drug: Bupivacaine (Block Drug)
  For block performances, 0,25% Bupivacaine will be used at 0,5 ml/kg (max. 20cc) for each side.
  Other Names: SPSIP Block
  Arms: SPSIPB Group

SUMMARY:
The aim is to compare the postoperative analgesic efficacy of serratus anterior plane block (SAPB) and serratus posterior superior intercostal plane block (SPSIPB) in patients undergoing mammoplasty surgery. To this end, a double-blind, randomized, controlled study has been designed. Female patients aged 18-65 years who will undergo mammoplasty surgery will be included in the study. Postoperative pain levels, opioid consumption, duration of analgesic requirement, and patient satisfaction will be evaluated in patients who receive fascial blocks for analgesic purposes.

DETAILED DESCRIPTION:
Pain management after breast surgery plays an important role in the patients' recovery process. Therefore, investigating effective and safe analgesic methods is important for improving patient comfort in the postoperative period. The serratus anterior plane block (SAPB) is a regional anesthesia technique commonly used for pain control after breast surgery. SAPB has been shown to be effective in reducing postoperative pain and decreasing opioid consumption. In addition, SAPB is easy to perform and has a low risk of complications. The serratus posterior superior intercostal plane block (SPSIPB) is a new technique developed to provide analgesia in thoracic surgeries. SPSIPB has been reported to be effective in reducing postoperative pain and decreasing analgesic consumption. However, data on the efficacy of SPSIPB in breast surgery are limited. This study aims to compare the postoperative analgesic efficacy of SAPB and SPSIPB in patients undergoing mammoplasty. For this purpose, a double-blind, randomized, controlled trial has been designed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years
* Patients undergoing elective mammoplasty
* ASA physical status I-II

Exclusion Criteria:

* Patients who refuse to participate
* Mentally disabled patients
* Presence of infection at the injection site
* Patients with coagulopathy
* History of allergy or toxicity to local anesthetics
* Patients with uncontrolled hypertension
* Patients with uncontrolled diabetes mellitus
* Patients with hepatic or renal failure
* Pregnant, breastfeeding women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females who are planned mammoplasty operation
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 0, 1, 6, 12 and 24 hours
  Tramadol will be prepared at a concentration of 10 mg/mL, and patient-controlled analgesia (PCA) will be administered without a basal infusion, using a lock-out interval of 20 minutes and a bolus dose of 20 mg.
Postoperative pain scores (Numerical rating scale: NRS),Between 0 and 10 points (11 points in total), as the score increases, the pain intensity increases. | 0, 1, 6, 12 and 24 hours
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 1, 6, 12 and 24 hours.

SECONDARY OUTCOMES:
Time to first analgesic requirement | 24 Hour
  Time from end of surgery to first analgesic requirement (min)
Patient satisfaction score | 24 Hour
  Overall patient satisfaction scores will be assessed using a 5-point Likert scale,Minimum value: 1, Maximum value: 5, where higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal Medical School, Bolu, Turkey (Türkiye)

REFERENCES:
- [Background] Koksal BG, Baytar C, Bayraktar E, Balbaloglu H. Effects of serratus posterior superior intercostal plane block on postoperative analgesia in patients undergoing breast cancer surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Apr 24;25(1):209. doi: 10.1186/s12871-025-03092-0. PMID 40275145